CLINICAL TRIAL: NCT06954207
Title: Analgesia for Total Hip Arthroplasty With PENG Block (ATHAPENG)
Acronym: ATHAPENG
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5166; 24-5166 (Other: HCL)
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Total Hip Arthroplasty for Osteoarthritis
Keywords: PENG block analgesia; Total hip arthroplasty; NOL index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient undergoing total hip arthroplasty for osteoarthritis under general anaesthesia with PENG blo: Patient undergoing total hip arthroplasty for osteoarthritis under general anaesthesia with PENG block
  Interventions: Device: Non interventional. Data collection concerns routine procedures and monitoring devices

INTERVENTIONS:
Device: Non interventional. Data collection concerns routine procedures and monitoring devices — Non interventional. Physiological parameters under general anesthesia are collected (arterial pressure, heart rhythm, bispectral index, NOL index, temperature, total dose of remifentanil infusion, analgesic drugs infusions). After surgery, pain scores (NRS), motor function and time to ambulation are also collected.

SUMMARY:
Analgesia for Total Hip Arthroplasty with PENG block (ATHAPENG)

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) for osteoarthritis is a commonly performed surgery worldwide. It is associated with significant pain, with median pain scores in the first 24 hours postoperatively exceeding 3 on the standardized numeric rating scale (NRS). Multimodal analgesia, including infusion of systemic analgesics and regional anesthesia through the Pericapsular Nerve Group Block (PENG block), has demonstrated efficacy in literature, when compared to other commonly used techniques such as the iliofascial block or surgical infiltration. However, analgesia provided by the PENG block appears to be incomplete, with a significant consumption of opioids in the postoperative period. The investigators hypothesis is that PENG block does not cover every hip sensitive territory involved during the surgical procedure.

The investigators conducted a single-center, observational, prospective study evaluating the antinociceptive effect of a PENG block performed preoperatively, at various surgical time points (incision, dislocation, femoral osteotomy, acetabular reaming, femoral reaming, femoral stem impaction, reduction, closure) by monitoring the Nociception Level Index (NOL index) during general anesthesia.

NOL index values (0 to 100) between 10 and 25 reflect nociception control, NOL index values exceeding 25 reflect excess of nociception, NOL index < 10 reflects a potential excess of opioids infusion.

After surgery, pain scores (NRS), opioid consumption, and the presence of motor blockade within the first 48 hours postoperatively were also assessed.

The aim of the study is to determine the efficacy of PENG block combined to multimodal analgesia on intraoperative nociception and postoperative pain in patients undergoing total hip arthroplasty under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years old)
* Undergoing primary hip arthroplasty for osteoarthritis
* Under general aneasthesia
* With PENG block

Exclusion Criteria:

* Patient under 18 years old
* Severe cognitive impairment or patient under guardianship
* Pregnancy
* Allergy to local anaesthetics
* Chronic pain with daily opioid consumption
* Non sinusal cardiac rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing scheduled total hip arthroplasty for osteoarthritis under general anaesthesia with PENG block.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Intraoperative nociception monitored by Nociception Level Index (NOL index) : mean and percentage of variations throughout surgery and within each surgical time points | NOL index is monitored in the operating room, during general anaesthesia while the surgical procedure is performed ( 60 to 120 minutes)
  To assess intra-operative nociception under general anaesthesia within each surgical time-points (incision, dislocation, femoral osteotomy, acetabular reaming, femoral reaming, femoral stem impaction, reduction, closure), NOL index is monitored continuously from anesthetic induction to end of surgery. Anaesthesiologist and nurse do not have access to the NOL screen monitor. Precise times of surgical time points are collected during surgery.
  Datas are then exported in excel files and investigators analyse:
  * Mean, median and max NOL index values during whole surgery
  * Mean, median and max NOL index values within each surgical time points
  * NOL index: percentage of time above values of 25 during whole surgery
  * NOL index : percentage of time above value of 25 within each surgical time points
  * Percentage of NOL variation within each time points

SECONDARY OUTCOMES:
Pain scores and opioid consumption | Day 0, day 1, day 2 postoperatively
  Pain scores evaluated by numeric rating scale (NRS, 0 to 10) are collected by nurses in charge of patients, in recovery room, and 6-12-24-48 hours postoperatively.
  Total dose of opioid consumption on day 1 and day 2 post operatively are collected through medical files.

CONTACTS AND LOCATIONS:
Locations (1):
- Edouard Herriot hospital, hospices civils de Lyon, Lyon, France